CLINICAL TRIAL: NCT04833361
Title: Pilot Evaluation of Potential Environmental Causes of Uveal Coloboma
Brief Title: Potential Environmental Causes of Uveal Coloboma
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000366; 000366-EI
Record Dates: First submitted 2021-04-05; First posted 2021-04-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09-30

CONDITIONS: Coloboma
Keywords: Questionnaire; Microphthalmia; Birth Defects; Natural History
MeSH Terms: conditions — Coloboma; Microphthalmos; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mothers: Mothers of children with coloboma.

SUMMARY:
Background:

Uveal coloboma is a congenital eye malformation. It is thought to be a genetic condition. But it might have environmental causes as well. Researchers want to study the mothers of children with coloboma. They will use parts of the National Birth Defects Prevention Study (NBDPS) Mother Questionnaire. NBDPS was a large study of birth defects. It collected data from 1997 to 2011. Researchers will use NBDPS and NIH data as well as the new survey to produce data that can serve as a basis for further study.

Objective:

To explore maternal factors and exposures during the first trimester of pregnancy as potential causes of uveal coloboma and to correlate exposure data to clinical data from affected children.

Eligibility:

Mothers of probands with coloboma who have taken part in NIH study 06-EI-0230, 04-EI-0039, or 13-EI-0049.

Design:

This is a hybrid study. It will use existing data from NBDPS and NIH studies. It will also use NBDPS for a new survey of mothers of children with coloboma.

Participants will take the survey by phone. Their pregnancy records may be reviewed. They will be asked about:

Important dates

Health and medicines

Tobacco, alcohol, and substance use

Parents occupations

Family demographics.

The survey will take 1 hour or less to complete.

Some data were obtained in past NIH studies. These data are largely from children. Some family data may be used as well. For example, eye exam data, gene test results, and family history of coloboma may be used. If a participant did not consent to the future use of their data, then their data will not be used.

Data will be stored in a secure NIH database.

...

DETAILED DESCRIPTION:
Study Description:

This evaluation of potential environmental causes of coloboma explores the experiences of a large cohort of mothers of children with uveal coloboma using portions of the National Birth Defects Prevention Study (NBDPS) Mother Questionnaire. It is postulated that maternal hypothyroidism and in utero alcohol exposure are found at higher rates in this cohort than in rates found in the general population. The goal is to produce descriptive statistic that could serve as a basis for further epidemiologic studies.

Objectives:

The primary objective is to explore maternal factors and exposures during the first trimester of pregnancy as potential causes of uveal coloboma and to correlate these exposures with the clinical presentation of the affected child/children.

ELIGIBILITY:
* INCLUSION CRITERIA:
* mothers of probands with coloboma that have previously been consented to an NIH protocol studying coloboma.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 180 mothers of probands with coloboma that have previously been consented to an NIH protocol studying coloboma.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
% of participants with x exposure compared to historical data | ongoing
  % of participants with x exposure compared to historical data from NBDPS study.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brooks, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided